CLINICAL TRIAL: NCT04205240
Title: Reduce Intensity Conditioning (RIC) Allogenic Hematopoietic Stem Cell Transplantation (Allo HSCT) for Patients With Relapsed Multiple Myeloma: A Pilot Study
Brief Title: Reduce Intensity Conditioning Donor Stem Cell Transplant for the Treatment of Relapsed Multiple Myeloma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Srinivas Devarakonda (Other)
Responsible Party: Sponsor-Investigator, Srinivas Devarakonda, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-19190; NCI-2019-07892 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-12-17; First posted 2019-12-19 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Recurrent Plasma Cell Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Stem Cell Transplantation; Cyclophosphamide; daratumumab; fludarabine; Melphalan; Mycophenolic Acid; Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (conditioning regimen, stem cell transplant) (Experimental): Patients receive fludarabine IV on days -5 to -2 and melphalan IV on days -3 to -2, then undergo stem cell transplantation on day 0. Patients receive cyclophosphamide on days 3 and 4, tacrolimus PO BID or IV starting on day 5, and mycophenolate mofetil IV or PO TID on days 5 to 35. Patients also receive daratumumab IV starting between days 90-150 for up to 1 year. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: Allogeneic Hematopoietic Stem Cell Transplantation; Drug: Cyclophosphamide; Biological: Daratumumab; Drug: Fludarabine; Drug: Melphalan; Drug: Mycophenolate Mofetil; Drug: Tacrolimus

INTERVENTIONS:
Procedure: Allogeneic Hematopoietic Stem Cell Transplantation — Undergo allogeneic hematopoietic stem cell transplantation
  Other Names: Allogeneic Hematopoietic Cell Transplantation; Allogeneic Stem Cell Transplantation; HSC; HSCT; Stem Cell Transplantation, Allogeneic
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamide Monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Biological: Daratumumab — Given IV
  Other Names: Anti-CD38 Monoclonal Antibody; Darzalex; HuMax-CD38; JNJ-54767414
Drug: Fludarabine — Given IV
  Other Names: Fluradosa
Drug: Melphalan — Given IV
  Other Names: Alanine Nitrogen Mustard; CB-3025; L-PAM; L-Phenylalanine mustard; L-Sarcolysin; L-Sarcolysin Phenylalanine mustard; L-Sarcolysine; Melphalanum; Phenylalanine Mustard; Phenylalanine Nitrogen Mustard; Sarcoclorin; Sarkolysin; WR-19813
Drug: Mycophenolate Mofetil — Given IV or PO
  Other Names: Cellcept; MMF
Drug: Tacrolimus — Given PO or IV
  Other Names: FK 506; Fujimycin; Hecoria; Prograf; Protopic

SUMMARY:
This phase II trial studies how well a reduced intensity conditioning regimen after donor stem cell transplant works in treating patients with multiple myeloma that has come back (relapsed). Drugs used in chemotherapy, such as cyclophosphamide, tacrolimus, and mycophenolate mofetil, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Immunotherapy with monoclonal antibodies, such as daratumumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving a reduce intensity conditioning regimen consisting of cyclophosphamide, tacrolimus, mycophenolate mofetil, and daratumumab after donor stem cell transplant may improve survival and reduce the risk of multiple myeloma coming back.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the 2-year progression-free survival (PFS) for haploidentical, matched or mismatched, related or unrelated reduce intensity allogenic hematopoietic stem cell transplantation (allo HSCT) in relapsed multiple myeloma (MM) patients.

SECONDARY OBJECTIVES:

I. To determine 2 year overall survival (OS). II. To determine the cumulative incidence of grade II-IV acute-graft-versushost-disease (aGVHD) at day 100 and 180.

III. To determine the 100 days, 1 year and 2 year cumulative incidence of treatment-related mortality (TRM).

IV. To assess one-year GVHD-free relapse-free survival (GRFS). V. To determine the cumulative incidence of chronic graft-versus-hostdisease (cGVHD) Va. To assess overall and best response rates 100 days after allo HCT, 3 months, 6 months and every 6 months thereafter until end of daratumumab maintenance.

VI. To determine rate of relapse after allo HSCT followed by maintenance. VII. To determine rate of minimal residual disease (MRD) negativity using next generation sequencing (Food and Drug Administration [FDA] approved) in patients achieving a very good partial response (VGPR) or better.

CORRELATIVE OBJECTIVE:

I. To determine immune reconstitution pattern on days +30, +100, +180 and +365 following allo HSCT.

OUTLINE:

Patients receive fludarabine intravenously (IV) on days -5 to -2 and melphalan IV on days -3 to -2, then undergo stem cell transplantation on day 0. Patients receive cyclophosphamide on days 3 and 4, tacrolimus orally (PO) or twice daily (BID) or IV starting on day 5, and mycophenolate mofetil IV or PO three times daily (TID) on days 5 to 35. Patients also receive daratumumab IV starting between day 90-150 for up to 1 year. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up periodically for up to 2 years post stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a partial response (PR) or better prior to allo-transplantation
* Relapsed MM with chemo sensitivity disease, with or without prior autologous HSCT
* First allogenic transplant
* Donors can be haploidentical, mismatch or matched related or unrelated. Stem cell source will be peripheral blood except for haploidentical where stem cell source will be bone marrow
* Ejection fraction >= 45%
* Estimated creatinine clearance greater than 40 mL/minute
* Diffusion capacity of the lung for carbon monoxide (DLCO) >= 40% (adjusted for hemoglobin)
* Forced expiratory volume in 1 second (FEV1) >= 50%
* Total bilirubin < 2 x the upper limit of normal
* Alanine aminotransferase (ALT)/aspartate aminotransferase (AST) < 2.5 x the upper normal limit
* Signed informed consent

Exclusion Criteria:

* Patients with polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin change (POEMS), Waldenstrom macroglobulinemia
* Uncontrolled bacterial, viral or fungal infection
* Patients with prior malignancies < 3 years except resected basal cell/squamous cell carcinoma, treated carcinoma in-situ. Other cancers treated with curative intent < 3 years previously will not be allowed unless approved by the principal investigator
* Female patients who are pregnant or breastfeeding. A negative pregnancy test will be required for all women of child bearing potential

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2021-05-08 (Actual); Study Completion 2021-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Srinivas Devarakonda, M.D., Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Conditioning Regimen, Stem Cell Transplant)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Conditioning Regimen, Stem Cell Transplant)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: 2-year Progression-free Survival (PFS)
Description: Patients who do not relapse or die will be censored at the date of last clinical assessment. Kaplan-Meier curves will be generated to estimate the PFS rates at 2 years posttransplant. To evaluate the potential association between patient characteristics and PFS, the log-rank test will be used to compare the PFS curves and Cox proportional hazard regression model will be used to estimate the hazard ratio.
Time Frame: From the date of transplant until the date of relapse or date of death from any cause, assessed at 2 years
Population: Due to low patient accrual to study unable to collect and analyze data
Arm/Group | Treatment (Conditioning Regimen, Stem Cell Transplant)
Number analyzed (Participants) | 0

2. Secondary Outcome: Incidence of Adverse Events
Description: Adverse events by grade will be summarized. The occurrence of grade 3+ adverse events according to Common Terminology Criteria for Adverse Events (CTCAE) will be summarized as well. Adverse events will initially be reviewed regardless of attribution, but also according to whether adverse events are possibly, probably, or definitely related to treatment.
Time Frame: Up to 2 years post-transplant
Population: Data was unable to be collected and analyzed due to low patient accrual to study
Arm/Group | Treatment (Conditioning Regimen, Stem Cell Transplant)
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Patients With Grade II-IV Acute Graft-versus Host Disease (GvHD (aGVHD)
Description: The event will be onset of grade II-IV aGvHD and time to aGvHD will be defined as the period of time from transplantation to the event of aGvHD. Death and early relapse without aGvHD will be competing risks. Cumulative incidence rate of aGVHD with 95% confidence intervals will be estimated from the cumulative incidence curves. To evaluate the association between patient characteristics and aGVHD, the Gray's test accounting for competing risks will be used to compare the cumulative incidence curves and a proportional hazards model for the sub distribution of competing risks will be used to estimate the hazard ratio. The cumulative incidence of chronic GVHD (cGVHD) will be similarly analyzed.
Time Frame: Up to 6 weeks
Measure: Number; unit: participants
Arm/Group | Treatment (Conditioning Regimen, Stem Cell Transplant)
Number analyzed (Participants) | 1
participants | 0

4. Secondary Outcome: Rate of Relapse
Description: Patients without relapse or death will be censored at last clinical assessment date. The similar analysis approach used for outcome of aGVHD will be applied.
Time Frame: From the date of transplant to relapse treating death from any cause as a competing risk, assessed up to 2 years
Population: Due to low patient accrual to study unable to collect and analyze data
Arm/Group | Treatment (Conditioning Regimen, Stem Cell Transplant)
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival (OS)
Description: A similar analysis approach described above for PFS will be applied for the OS analysis.
Time Frame: From the date of transplant to death or last contact date if no death, assessed up to 2 years
Population: Due to low patient accrual to study unable to collect and analyze data
Arm/Group | Treatment (Conditioning Regimen, Stem Cell Transplant)
Number analyzed (Participants) | 0

6. Secondary Outcome: 1- Year GVHD-free Relapse-free Survival (GRFS)
Description: Patients who do not experience an event will be censored at the date of last clinical assessment. A similar analysis approach described above for PFS will be applied for the GRFS analysis.
Time Frame: From the date of transplant until the date of grade II-IV acute GVHD, chronic GVHD, disease relapse or progression, or death from any cause, whichever occurs first, assessed at 1 year
Population: Due to low patient accrual to study unable to collect and analyze data
Arm/Group | Treatment (Conditioning Regimen, Stem Cell Transplant)
Number analyzed (Participants) | 0

7. Secondary Outcome: 100-day Cumulative Incidence of Treatment-related Mortality (TRM)
Description: The event will be death due to reasons other than disease. The competing risk for non relapsed mortality (NRM) will be death due to disease. The cumulative incidence curve accounting competing risks will be generated to estimate the cumulative incidence rate at various time points.
Time Frame: From the date of transplant to date of death, assessed up to 100 days
Population: Due to low patient accrual to study unable to collect and analyze data
Arm/Group | Treatment (Conditioning Regimen, Stem Cell Transplant)
Number analyzed (Participants) | 0

8. Secondary Outcome: 1-year Cumulative Incidence TRM
Description: The event will be death due to reasons other than disease. The competing risk for NRM will be death due to disease. The cumulative incidence curve accounting competing risks will be generated to estimate the cumulative incidence rate at various time points.
Time Frame: From the date of transplant to date of death, assessed at 1 year
Population: Due to low patient accrual to study unable to collect and analyze data
Arm/Group | Treatment (Conditioning Regimen, Stem Cell Transplant)
Number analyzed (Participants) | 0

9. Secondary Outcome: 2-year Cumulative Incidence of TRM
Description: as for outcome 8
Time Frame: From the date of transplant to date of death, assessed at 2 years
Population: Due to low patient accrual to study unable to collect and analyze data
Arm/Group | Treatment (Conditioning Regimen, Stem Cell Transplant)
Number analyzed (Participants) | 0

10. Secondary Outcome: Overall Response Rate
Description: The proportion of each type of response with a 95% confidence interval (CI) will be reported for all evaluable patients, assuming a binomial distribution.
Time Frame: Up to 2 years post-transplant
Population: Due to low patient accrual to study unable to collect and analyze data
Arm/Group | Treatment (Conditioning Regimen, Stem Cell Transplant)
Number analyzed (Participants) | 0

11. Secondary Outcome: Number of Patients With a Partial Response
Description: The proportion of each type of response with a 95% CI will be reported for all evaluable patients, assuming a binomial distribution.
Time Frame: Approximately 11 months
Measure: Number; unit: patients
Arm/Group | Treatment (Conditioning Regimen, Stem Cell Transplant)
Number analyzed (Participants) | 1
patients | 1

12. Other Pre Specified Outcome: Rate of Minimal Residual Disease-negativity
Description: Will be defined as the proportion of patients who achieved minimal residual disease-negative status at the respective time point, in accordance with the International Myeloma Working Group criteria. Minimal residual disease was evaluated by next-generation sequencing using ClonoSEQ Assay.
Time Frame: Baseline up to 365 days post-transplant
Population: Due to low patient accrual to study unable to collect and analyze data
Arm/Group | Treatment (Conditioning Regimen, Stem Cell Transplant)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event information was collected for patients from baseline through study completion utilizing the CTCAE version 5.0 to determine the severity of the reaction for adverse event reporting from baseline to after study completion up to 1 year.
Arm/Group | Treatment (Conditioning Regimen, Stem Cell Transplant)
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Conditioning Regimen, Stem Cell Transplant) (N=1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Metabolism and Nutrition Disorders (Metabolism and nutrition disorders) | 1 (1)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Conditioning Regimen, Stem Cell Transplant) (N=1)
Abdominal Distension (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Alkaline phosphatase increased (Investigations) | 1 (1)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bronchial stricture (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Chronic Kidney Disease (Renal and urinary disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epstein-Barr virus infection reactivation (Infections and infestations) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Forced expiratory volume decreased (Investigations) | 1 (1)
Generalized edema (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Hallucinations (Psychiatric disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial was terminated early due to poor patient accrual

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/40/NCT04205240/Prot_SAP_002.pdf
  • Informed Consent Form (2021-03-11): https://cdn.clinicaltrials.gov/large-docs/40/NCT04205240/ICF_003.pdf